CLINICAL TRIAL: NCT02585180
Title: Subglottic Secretions Surveillance to Predict Bacterial Pathogens Involved in Ventilator-associated Pneumonia (VAP): an Ancillary Study of the DEMETER Trial (NCT02515617)
Brief Title: Subglottic Secretions Surveillance to Predict Bacterial Pathogens Involved in Ventilator-associated Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Collaborators: Ministry of Health, France (Other Government); University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CHD 052-15
Record Dates: First submitted 2015-10-20; First posted 2015-10-23 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Ventilator-associated Pneumonia
Keywords: Ventilator-associated pneumonia; Surveillance; Subglottic-secretions; Critically ill patients; Prevention
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Period with endotracheal tubes not allowing SSD (Active Comparator): During this period of the DEMETER study (NCT02515617), patients will be intubated with standard endotracheal tubes not allowing Subglottic Secretions Drainage
  Interventions: Device: Endotracheal tubes not allowing SSD
- Period with endotracheal tubes allowing SSD (Experimental): During this period of the DEMETER study (NCT02515617), patients will be intubated with specific endotracheal tubes allowing Subglottic Secretions Drainage
  Interventions: Device: Endotracheal tubes allowing SSD

INTERVENTIONS:
Device: Endotracheal tubes not allowing SSD — In each participating center, a bundle of VAP prevention will be applied: elevate the head of the bed to 30°-45°, regular oral care, manage patients with sedation algorithm, assess readiness to extubate daily, intermittent control of endotracheal tube cuff pressure
  Arms: Period with endotracheal tubes not allowing SSD
Device: Endotracheal tubes allowing SSD — In each participating center, a bundle of VAP prevention will be applied: elevate the head of the bed to 30°-45°, regular oral care, manage patients with sedation algorithm, assess readiness to extubate daily, intermittent control of endotracheal tube cuff pressure.
  In addition, SSD will be realized using a 10 ml syringe at in attending frequency of 2 hours.
  Arms: Period with endotracheal tubes allowing SSD

SUMMARY:
Many studies provide evidence for the benefit of lower respiratory tract surveillance, mostly by culture of endotracheal secretions, to predict bacterial pathogens (especially multi-drugs resistant pathogens) involved in VAP. The DEMETER study (NCT02515617) assessing the medico-economical impact of the subglottic secretions drainage (SSD) provides the opportunity to evaluate the accuracy of the subglottic secretions culture surveillance to predict pathogens involved in VAP (in comparison with the concomitant endotracheal secretions surveillance). These subglottic and tracheal secretions culture surveillance will be masked to the investigators of the DEMETER Study.

This ancillary study will be performed in 14 centers participating to the DEMETER study

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Invasive mechanical ventilation delivered via an endotracheal tube and expected to be required more than 24 hours
* Intubation performed in units in which the specific endotracheal tube allowing the subglottic secretions drainage will be available during the SSD period of the trial
* Information delivered

Exclusion Criteria:

* Previous inclusion in the study
* Patients moribund at the Intensive Care Unit admission
* Pregnant, parturient or breast-feeding woman
* Patient hospitalized without consent and/or deprived of liberty by court's decision
* Patient under guardianship or curators
* Lack of social insurance
* Concomitant inclusion in a trial on VAP prevention
* Patient with no comprehension of the French language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2015-11-04 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
Rate of adjudicated VAP in which the bacteria involved have been, previously, detected with the subglottic secretions culture surveillance. | Until weaning of mechanical ventilation, an expected average of 10 days
  For each episode of VAP, bacteria involved will be compared with bacteria isolated, previously, into the subglottic secretions. This comparison will be performed by the microbiologist of each center. A bacteria isolated into the subglottic secretions will be considered as the same than the one involved in VAP if these 2 same micro-organisms have the same antibiotics susceptibility. Moreover, for the comparison, the third last subglottic secretions samples, if available, obtained before the VAP occurrence, will be taking account.

SECONDARY OUTCOMES:
Rate of adjudicated VAP in which the bacteria involved have been, previously, detected with the tracheal secretions culture surveillance. | Until weaning of mechanical ventilation, an expected average of 10 days
  For each episode of VAP, bacteria involved will be compared with bacteria isolated, previously, into the tracheal secretions. This comparison will be performed by the microbiologist of each center. A bacteria isolated into the tracheal secretions will be considered as the same than the one involved in VAP if these 2 same microorganisms have the same antibiotics susceptibility. Moreover, for the comparison, the third last tracheal secretions samples, if available, obtained before the VAP occurrence will be taking account.
Adequate probabilistic antibiotherapy initiated during the study by the investigators in case of adjudicated VAP | Until weaning of mechanical ventilation, an expected average of 10 days
  Proportion of VAP for whom the probabilistic antibiotherapy used during the trial appeared to be empirically active
Adequate theoretical probabilistic antibiotherapy with the knowledge of the subglottic culture surveillance | Until weaning of mechanical ventilation, an expected average of 10 days
  Proportion of adjudicated VAP for whom a theoretical probabilistic antibiotherapy would be empirically active with the knowledge of the results of the subglottic secretions samples obtained more than 3 days before the occurrence of VAP. The theoretical antibiotherapy will be determined by an independent committee unaware of the type of samples evaluated (subglottic or tracheal secretions).
Adequate theoretical probabilistic antibiotherapy with the knowledge of the tracheal culture surveillance | Until weaning of mechanical ventilation, an expected average of 10 days
  Proportion of adjudicated VAP for whom a theoretical probabilistic antibiotherapy would be empirically active with the knowledge of the results of the tracheal secretions samples obtained more than 3 days before the occurrence of VAP. The theoretical antibiotherapy will be determined by an independent committee unaware of the type of samples evaluated (subglottic or tracheal secretions).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude LACHERADE, MD, Principal Investigator — CHD VENDEE
Locations (15):
- CHU André Vésale, Montigny-le-Tilleul, Belgium
- France (14):
  - CH Annecy Genevois, Annecy
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - Centre Hospitalier Intercommunal des Portes de l'Oise, Beaumont-sur-Oise
  - Chd Vendee, La Roche-sur-Yon
  - CH Docteur Schaffner, Lens
  - CH de Montauban, Montauban
  - Centre Hospitalier Régional d'Orléans, Orléans
  - CHU Pointe à Pitre les Abymes, Pointe à Pitre
  - CHI Poissy Saint Germain, Poissy
  - Centre Hospitalier René Dubos, Pontoise
  - CHU La Réunion, site de Saint Denis de la Réunion, Saint-Denis (Réunion)
  - CH de Saint Nazaire, Saint-Nazaire
  - CHU de Strasbourg Nouvel Hôpital Civil, Strasbourg
  - CHU Tours, site Bretonneau, Tours

REFERENCES:
- [Background] Brusselaers N, Labeau S, Vogelaers D, Blot S. Value of lower respiratory tract surveillance cultures to predict bacterial pathogens in ventilator-associated pneumonia: systematic review and diagnostic test accuracy meta-analysis. Intensive Care Med. 2013 Mar;39(3):365-75. doi: 10.1007/s00134-012-2759-x. Epub 2012 Nov 28. PMID 23188467